CLINICAL TRIAL: NCT03634215
Title: Estimation of Coagulation Factor XIII Activity Based on the Initial Plasma Fibrinogen Level in Trauma
Status: Completed | Type: Observational
Sponsor: Masaryk Hospital Krajská zdravotní a.s. (Other)
Responsible Party: Principal Investigator, Josef Skola, Clinical Director, Masaryk Hospital Krajská zdravotní a.s.
Other Study IDs: KAPIM-2
Record Dates: First submitted 2018-07-01; First posted 2018-08-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Multiple Trauma; Coagulation Disorder; Coagulation Factor Deficiency; Coagulation Defect; Acquired
MeSH Terms: conditions — Multiple Trauma; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Trauma patients
  Interventions: Diagnostic Test: fibrinogen plasma concentration, coagulation factor XIII activity

INTERVENTIONS:
Diagnostic Test: fibrinogen plasma concentration, coagulation factor XIII activity — blood sampling for a routine coagulation test

SUMMARY:
Coagulation factor XIII (FXIII), a plasma transglutaminase, is known as the final enzyme of the coagulation cascade, responsible for a cross-linking of fibrin to strengthen blood clot. It also minimizes fibrin degradation by its cross-linking it with alfa2-antiplasmin molecules. It has been found that similar to plasma fibrinogen level, FXIII activity can be reduced in the early phase of severe trauma. Therefore, its immediate substitution is of potential therapeutic interest in trauma-induced coagulopathy. However, unlike plasma fibrinogen level evaluation, measurement of the FXIII activity is not routinely available. Therefore, targeted substitution of FXIII is practically impossible. The plasma fibrinogen level is routinely measured in severe trauma patients. Based on pathophysiologic assumptions and a limited number of published data we hypothesize that the FXIII activity correlates with fibrinogen level. In such case, indirect FXIII activity prediction by fibrinogen level measurement would be a convenient approach to enable FXIII targeted substitution. Therefore we decided to perform a prospective observational clinical trial to determine whether the low plasma fibrinogen level in severe trauma correlates with decreased FXIII activity.

DETAILED DESCRIPTION:
Coagulation factor XIII (FXIII), a plasma transglutaminase, is known as the final enzyme of the coagulation cascade, responsible for a cross-linking of fibrin to strengthen blood clot. It also minimizes fibrin degradation by its cross-linking it with alfa2-antiplasmin molecules. It has been found that similar to plasma fibrinogen level, FXIII activity can be reduced in the early phase of severe trauma. Therefore, its immediate substitution is of potential therapeutic interest in trauma-induced coagulopathy. However, unlike plasma fibrinogen level evaluation, measurement of the FXIII activity is not routinely available. Therefore, targeted substitution of FXIII is practically impossible. The plasma fibrinogen level is routinely measured in severe trauma patients. Based on pathophysiologic assumptions and a limited number of published data we hypothesize that the FXIII activity correlates with fibrinogen level. In such case, indirect FXIII activity prediction by fibrinogen level measurement would be a convenient approach to enable FXIII targeted substitution. Therefore we decided to perform a prospective observational clinical trial to determine whether the low plasma fibrinogen level in severe trauma correlates with decreased FXIII activity.

ELIGIBILITY:
Inclusion Criteria:

* a patient with presumed severe trauma admitted to the participating centre

Exclusion Criteria:

* inflammatory disease
* malignant disease
* pregnancy
* receipt of any fibrinogen / coagulation factor XIII product before blood sampling
* patients on dabigatran

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with presumed severe trauma as assessed by the national trauma triage criteria admitted to a participating centre.
Sampling Method: Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
coagulation factor XIII activity | 1 day
  coagulation factor XIII activity expressed as % of the normal value

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - Krajska nemocnice Liberec, Liberec, Liberecký kraj
  - Fakultní nemocnice Plzen, Pilsen, Plzeň Region
  - Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem, Ústecký kraj

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dickneite G, Herwald H, Korte W, Allanore Y, Denton CP, Matucci Cerinic M. Coagulation factor XIII: a multifunctional transglutaminase with clinical potential in a range of conditions. Thromb Haemost. 2015 Apr;113(4):686-97. doi: 10.1160/TH14-07-0625. Epub 2015 Feb 5. PMID 25652913
- [Background] Theusinger OM, Baulig W, Seifert B, Muller SM, Mariotti S, Spahn DR. Changes in coagulation in standard laboratory tests and ROTEM in trauma patients between on-scene and arrival in the emergency department. Anesth Analg. 2015 Mar;120(3):627-635. doi: 10.1213/ANE.0000000000000561. PMID 25545751
- [Background] Sorensen B, Fries D. Emerging treatment strategies for trauma-induced coagulopathy. Br J Surg. 2012 Jan;99 Suppl 1:40-50. doi: 10.1002/bjs.7770. PMID 22441854